CLINICAL TRIAL: NCT04140942
Title: Improving Employment and Reducing Recidivism Among Prison Offenders Via Virtual Interview Training Tool (MICHR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Matthew Smith, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00165245; 3UL1TR002240-05S1 (NIH)
Record Dates: First submitted 2019-10-23; First posted 2019-10-28 (Actual); Results first posted 2023-03-30 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Criminal Behavior
MeSH Terms: conditions — Criminal Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Services as usual + Virtual Reality Job Interview Training (Experimental): In addition to the services as usual, participants will participate in Virtual Reality Job Interview Training.
  Interventions: Behavioral: Virtual Reality Job Interview Training; Behavioral: Services as usual
- Services as Usual (Active Comparator): Study participants will be receiving their Vocational Village services as usual that may include but not limited to vocational skill training, and social skill training.
  Interventions: Behavioral: Services as usual

INTERVENTIONS:
Behavioral: Virtual Reality Job Interview Training — Participants will engage in training related to preforming well during a job interview as well as repeated job interview practice with a virtual hiring manager. Participants will receive feedback and tips on improving skills throughout training.
  Arms: Services as usual + Virtual Reality Job Interview Training
Behavioral: Services as usual — Study participants will be receiving Vocational Village services as usual that may include but is not limited to vocational skill training, daily living skill training, and social skill training.

SUMMARY:
The goal is to conduct a feasibility effectiveness RCT of Virtual Interview Training (VIT) by comparing employment and recidivism outcomes of offenders (25 years and older) receiving vocational services as usual (SAU) plus VIT (SAU+VIT) with the outcomes of offenders receiving only services as usual (SAU-only).

The plan calls for participants to include offenders who are at moderate to high risk for reoffending (with an emphasis on violent-crime reoffending) who are currently enrolled in a Vocational Village Prison Setting with the Michigan Department of Corrections.

DETAILED DESCRIPTION:
More than 600,000 ex-offenders re-enter the community from prison each year and 50% of them recidivate within 12 months of release. Employment significantly reduces the risk of recidivism for ex-offenders, and as such, is a critical target for intervention. However, evidence-based employment services are rarely delivered in prisons. Moreover, employment services that are available do not include evidence-based job interview training. Virtual Reality Job Interview Training (VR-JIT) is an evidence-based tool that was developed and evaluated with funding from the National Institute of Mental Health. However, VR-JIT has a feature to practice discussing a prior conviction during a job interview that has not yet been evaluated. Given that an ex-offender's job interview outcome may depend on discussing their prior conviction, we are partnering with the Michigan Department of Corrections (MDOC) to evaluate if delivering VR-JIT within their Vocational Village program can improve employment and reduce recidivism among offenders after their release from prison. Thus, there are two goals for this pilot study. We will evaluate the preliminary effectiveness of whether VR-JIT added to Vocational Village services-as-usual improves outcomes (interview skills, employment, recidivism) for offenders after their release from prison (at a 6-month follow-up visit). These preliminary data will support a proposal to a federal agency for a fully-powered randomized controlled trial to evaluate the effectiveness of VR-JIT with prison settings.

ELIGIBILITY:
Inclusion Criteria:

* 25 years or older
* Identified as at moderate to high risk for reoffending with violent crimes (determined at the time of enrollment in the Vocational Village via the COMPAS Risk Assessment Classification Instrument [60])
* Within three months of their earliest release date
* Actively enrolled in a Vocational Village
* Have at least a 6th grade reading comprehension

Exclusion Criteria:

* Has uncorrected hearing or visual problem that prevents him or her from using the training
* Has a medical illness that compromises their cognition (for example, moderate to severe traumatic brain injury).

Min Age: 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Smith, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Services as Usual | Services as Usual + Virtual Reality Job Interview Training
Started | 16 | 28
Completed Post Test Only (Reason for incompletion of post test included: COVID-19 shutdown, early release from prison, and drop out.) | 11 | 22
Completed (Included in employment analysis) | 16 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Services as Usual | Services as Usual + Virtual Reality Job Interview Training | Total
Number analyzed (Participants) | 16 | 28 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (8.9) | 38.1 (6.1) | 38.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 28 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 9 | 13 | 22
  White | 6 | 13 | 19
  LatinX | 0 | 2 | 2
  More than one race | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 28 | 44
Current Grade [Count of Participants; unit: Participants]
  High school graduate/GED equivalent | 7 | 13 | 20
  Some college | 5 | 4 | 9
  Technical school graduate | 4 | 9 | 13
  Associate's degree | 0 | 2 | 2
Prior Employment [Count of Participants; unit: Participants] | 15 | 27 | 42
Psychological Distress - DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure - Adult [Mean (Standard Deviation); unit: units on a scale] — The DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure - Adult is a self rated measure that assesses mental health domains with 23 questions. For this study, we excluded Suicidal Ideation and two Substance Use questions, so our total scale was 21. Items are on a 5-point scale (0 = none or not at all; 1 = slight or rare, less than a day or two; 2 = mild or several days; 3 = moderate or more than half the days; and 4 = severe or nearly every day). Scores can range from 0 to 84. A higher score represents a more severe/negative outcome of higher psychological distress.
  units on a scale | 3.7 (6.1) | 2.1 (3.3) | 2.7 (4.5)
Self-reported Mental Health Disorders [Count of Participants; unit: Participants]
  Depressive disorder | 4 | 5 | 9
  Anxiety disorder | 4 | 2 | 6
  Bipolar disorder | 3 | 2 | 5
  Posttraumatic stress disorder | 2 | 2 | 4
Risk for Non-Violent Reoffense [Count of Participants; unit: Participants] — Risk for Non-Violent Reoffense is a component of the Correctional Offender Management Profiling for Alternative Sanctions tool, commonly known as COMPAS, for criminogenic risk and needs assessments and unified case planning. Scores were obtained from MDOC staff and the scores indicate Low, Medium, and High risk for non-violent re-offense.
  Participants
    Medium | 7 | 13 | 20
    High | 9 | 15 | 24
Risk for Violent Reoffense [Count of Participants; unit: Participants]
  Medium | 8 | 17 | 25
  High | 8 | 11 | 19
Criminal Justice History: Arrest Count [Mean (Standard Deviation); unit: count] — Arrest count was a self-reported measure of how many times a participant had been arrested. Higher counts indicated more times arrested.
  count | 8.3 (9.4) | 8 (4.9) | 8.1 (6.8)
Criminal Justice History: Total Years in Prison/Jail [Mean (Standard Deviation); unit: years] — Total Years in Prison/Jail was a self-reported question asking participants how many years they spent in prison/jail. Higher numbers indicated a higher time spent in prison/jail.
  years | 8.8 (6.6) | 6.3 (4.2) | 7.2 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Employment as Measured in Outcome Questionnaire
Description: Employment rate will be measured by participant self-report using a questionnaire.
Time Frame: 6 Month & 12 month follow up after villagers are released.
Measure: Count of Participants; unit: Participants
Arm/Group | Services as Usual | Services as Usual + Virtual Reality Job Interview Training
Number analyzed (Participants) | 16 | 28
Participants
  6-Month Employment | 11 | 23
  12-Month Employment | 14 | 24
Statistical Analysis 1: Comparison: Services as Usual vs Services as Usual + Virtual Reality Job Interview Training; 6-Month Employment; Test type: Superiority; p = .15, Chi-squared
Statistical Analysis 2: Comparison: Services as Usual vs Services as Usual + Virtual Reality Job Interview Training; 6-Month Employment; Test type: Superiority; p = .001, Regression, Logistic
Statistical Analysis 3: Comparison: Services as Usual vs Services as Usual + Virtual Reality Job Interview Training; 12-Month Employment; Test type: Superiority; p = .87, Chi-squared

2. Primary Outcome: Job Interview Skills From Mock Interview Rating Scale (MIRS)
Description: Interviewing skills were measured using a role-play measure in which subjects act out two job interview scenarios with trained actors. Interviews were video recorded and scored. An average of the two scenarios at baseline was used to create a single pretest score and an average of the two scenarios at posttest was used to create a single posttest score. The method of assessment is the job interview skills rating scale as measured by the Mock Interview Rating Scale (MIRS). Possible scores range from 8 to 40, with higher scores indicating better interview skills.
Time Frame: Pretest (Baseline) and Posttest (approximately 6 weeks after Baseline)
Population: Those not included in analysis were for the following reasons: missing post-test data (n=11), inaudible study data (n=2), administratively withdrawn due self-disclosed anxiety about failing to be released from prison (n=1). n=6 excluded from SAU and n=8 excluded from SAU+VR-JIT.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Services as Usual | Services as Usual + Virtual Reality Job Interview Training
Number analyzed (Participants) | 10 | 20
score on a scale
  Pretest score | 31.8 (2.3) | 29.9 (1.5)
  Posttest score | 31.6 (1.7) | 33.2 (1.1)
Statistical Analysis 1: Comparison: Services as Usual vs Services as Usual + Virtual Reality Job Interview Training; Test type: Superiority; p = 0.04, ANCOVA; Repeated measures

3. Primary Outcome: Number of Participants on With at Least 1 Yes Answer to Recidivism Self-Report Questionnaire
Description: Recidivism status will be collected via follow up self-report survey with a questions asking if they have been re-arrested (yes/no). The recidivism self-report data will be validated by administrative data collected from MDOC.
Time Frame: 6 Month and 12 months after Villager Release Date
Measure: Count of Participants; unit: Participants
Arm/Group | Services as Usual | Services as Usual + Virtual Reality Job Interview Training
Number analyzed (Participants) | 16 | 28
Participants
  Number of Participants Re-Arrested within 6-Months after their Release Date | 1 | 0
  Number of Participants Re-Arrested within 12-Months after their Release Date | 1 | 0
Statistical Analysis 1: Comparison: Services as Usual vs Services as Usual + Virtual Reality Job Interview Training; 12-Month Recidivism Analysis; Test type: Superiority; p = .056, Chi-squared
Statistical Analysis 2: Comparison: Services as Usual vs Services as Usual + Virtual Reality Job Interview Training; 6-Month Recidivism Analysis; Test type: Superiority; p = .18, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse Event data were monitored/assessed through study completion (an average of 1 year per participant)
Arm/Group | Services as Usual | Services as Usual + Virtual Reality Job Interview Training
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/28
Other Adverse Events (participants affected / at risk) | 0/16 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-06-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT04140942/Prot_SAP_000.pdf
  • Informed Consent Form: In-Person Consent (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT04140942/ICF_001.pdf
  • Informed Consent Form: Virtual Consent (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT04140942/ICF_002.pdf